CLINICAL TRIAL: NCT06339034
Title: Repurposing Lithium as a Disease-modifying Therapy in Parkinson's Disease: A Randomized Controlled Trial
Brief Title: Repurposing Lithium for Parkinson's Disease: a RCT
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Cure Parkinson's (Other)
Responsible Party: Principal Investigator, Thomas Guttuso, Professor of Neurology, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY
Record Dates: First submitted 2024-03-24; First posted 2024-04-01 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson's; Lithium; Free water; Disease-modifying therapy
MeSH Terms: conditions — Parkinson Disease | interventions — Lithium

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lithium (Active Comparator): Lithium: 10mg, 2x/day
  Interventions: Dietary Supplement: Lithium
- Placebo (Placebo Comparator): Identical capsules filled with cellulose: 10mg, 2x/day
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lithium — 5mg of elemental lithium/capsule
  Arms: Lithium
Other: Placebo — Cellulose-filled capsules
  Arms: Placebo

SUMMARY:
This study will examine the effects of lithium 20mg/day compared to placebo on MRI and blood-based biomarkers among 20 early-stage Parkinson's disease patients.

DETAILED DESCRIPTION:
In observational studies, small daily doses of lithium have been associated with a 77% reduced risk of developing Parkinson's disease (PD). In addition, lithium therapy has been effective in preventing neuronal death and behavioral symptoms in several PD animal models. Recently, our group has shown 24-weeks of low-dose lithium therapy in PD to improve both MRI and blood-based biomarkers implying that lithium may be slowing the progression of the disease. However, these findings stem from only three of four patients receiving MRIs. A larger study will be required to determine if these promising results can be replicated. The proposed study will enroll 20 additional PD patients who will be randomly assigned to receive either lithium 20mg/day or identically-appearing placebo capsules for 24 weeks. This will be a double-blind study meaning that neither the patients nor the study team will know to which therapy patients have been assigned. Positive results from this study will support further research on lithium that could eventually support lithium as a disease-modifying therapy for PD that could improve patients' long-term prognoses.

ELIGIBILITY:
Inclusion Criteria:

* Have PD for <4 years diagnosed by a movement disorder specialist. Have normal thyroid and renal function at the screening visit. Have no previous exposure to lithium therapy. Have no history of brain surgery. Have no hx of brain imaging findings suggesting another neurological condition besides PD.

Have no use of tobacco or THC products for >1 year. Have stable PD medications for >30 days without current need for adjustments in the investigator's opinion.

Have stable psychiatric and diuretic medications for >60 days with no anticipated need for changes for at least 24 weeks.

Have no active medical or psychiatric condition that may interfere with study procedures in the investigator's opinion.

Exclusion Criteria:

* Have PD for >4 years or does not have PD. Have abnormal normal thyroid and renal function at the screening visit. Have previous exposure to lithium therapy. Have history of brain surgery. Have hx of brain imaging findings suggesting another neurological condition besides PD.

Have use of tobacco or THC products within the past year. Have PD medication adjustments within 30 days or needs PD medication adjustments in the investigator's opinion.

Have psychiatric or diuretic medication adjustments within the last 60 days or is anticipated to need changes over next 24 weeks.

Have active medical or psychiatric condition that may interfere with study procedures in the investigator's opinion.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
MRI-derived free water (FW) levels. | Change from baseline (BL) to 24 week
  FW in the posterior substantia nigra (pSN), dorsomedial nucleus of the thalamus (DMN-T) and the nucleus basalts of Meynert (nbM).
Peripheral blood mononuclear cell (PBMC) nuclear receptor-related 1 protein (Nurr1) mRNA expression | Change from baseline (BL) to 24 week
  PBMC Nurr1 mRNA expression using Taqman PCR.
Serum neurofilament light chain (NfL) | Change from baseline (BL) to 24 week
  Serum NfL assessed using SIMOA platform by Quanterix (Lexington, MA)

SECONDARY OUTCOMES:
PBMC superoxide dismutase type-1 (SOD-1) mRNA expression | Change from baseline (BL) to 24 week
  PBMC SOD-1 mRNA expression using Taqman PCR
PBMC pS9/total glycogen synthase kinase-3B (GSK-3B) ratio | Change from baseline (BL) to 24 week
  Assessed using ELISA
PBMC pThr308 and pS473/total protein kinase B (Akt) ratios | Change from baseline (BL) to 24 week
  Assessed using ELISA
Serum interleukin-6 | Change from baseline (BL) to 24 week
  Assessed using ELISA
Serum glial fibrillary acidic protein (GFAP) | Change from baseline (BL) to 24 week
  Serum GFAP assessed using SIMOA platform by Quanterix (Lexington, MA)
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III (Motor Examination) | Change from baseline (BL) to 24 week
  Assessed in the "on" state. Score range 0-132 with higher scores indicating worse outcomes.
Montreal Cognitive Assessment (MoCA) | Change from baseline (BL) to 24 week
  Score range 0-30 with higher scores indicating better outcomes.
Parkinson's Anxiety Scale | Change from baseline (BL) to 24 week
  Score range 0-48 with higher scores indicating worse outcomes.
Geriatric Depression Scale-15 | Change from baseline (BL) to 24 week
  Score range 0-15 with higher scores indicating worse outcomes.
Fatigue Severity Scale | Change from baseline (BL) to 24 week
  Score range 9-63 with higher scores indicating worse outcomes.
Insomnia Severity Index | Change from baseline (BL) to 24 week
  Score range 0-28 with higher scores indicating worse outcomes.
Parkinson's Disease Questionnaire-8 | Change from baseline (BL) to 24 week
  Score range 0-32 with higher scores indicating worse outcomes.
Levodopa equivalent daily dose (LEDD) | Change from baseline (BL) to 24 week
  Higher scores indicate higher dose of dopaminergic therapy.

OTHER OUTCOMES:
Adverse events | Throughout 24 week study
  Number of patients with any and serious adverse events and number who withdraw from the study.

CONTACTS AND LOCATIONS:
Locations (1):
- UBMD Neurology, Williamsville, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will be considered on a case-by-case basis.

REFERENCES:
- [Background] Guttuso T Jr, Shepherd R, Frick L, Feltri ML, Frerichs V, Ramanathan M, Zivadinov R, Bergsland N. Lithium's effects on therapeutic targets and MRI biomarkers in Parkinson's disease: A pilot clinical trial. IBRO Neurosci Rep. 2023 May 7;14:429-434. doi: 10.1016/j.ibneur.2023.05.001. eCollection 2023 Jun. PMID 37215748